CLINICAL TRIAL: NCT00439517
Title: A Randomized, Open-label Phase II Study Evaluating the Efficacy and Safety of FOLFOX-4 Plus Cetuximab Versus UFOX Plus Cetuximab as First-line Therapy in Subjects With Metastatic Colorectal Cancer.
Brief Title: Study to Evaluate the Efficacy and Safety of FOLFOX-4 Plus Cetuximab Versus UFOX Plus Cetuximab.
Acronym: FUTURE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMR200025-001
Record Dates: First submitted 2007-02-22; First posted 2007-02-23 (Estimated); Results first posted 2011-06-14 (Estimated); Last update posted 2014-06-27 (Estimated); Status verified 2014-06

CONDITIONS: Previously Untreated Metastatic Colorectal Cancer
Keywords: Cancer; Colorectal; Metastatic; Untreated
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis | interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): UFOX + Cetuximab
  Interventions: Drug: UFOX + Cetuximab
- 2 (Active Comparator): FOLFOX4 + Cetuximab
  Interventions: Drug: FOLFOX4 + Cetuximab

INTERVENTIONS:
Drug: UFOX + Cetuximab — * Cetuximab infusion (400 mg/m^2 on day 1 of cycle 1 and 250 mg/m^2 at each subsequent day 1, as well as on days 8, 15 and 22)
  * Oxaliplatin infusion (85mg/m^2) on days 1 and 15 (every 2 weeks)
  * Oral UFT® (250mg/m^2 tegafur + 560 mg/m^2 uracil in 3 daily doses rounded to the nearest number of whole capsules) on days 1-21
  * Oral Folinic Acid (90 mg in 3 daily divided doses) on days 1-21
  Arms: 1
Drug: FOLFOX4 + Cetuximab — * Cetuximab infusion (400 mg/m^2 on day 1 of cycle 1 and 250 mg/m^2 at each subsequent day 1, as well as on days 8, 15 and 22)
  * Oxaliplatin infusion (85 mg/m^2) on days 1 and 15 (every 2 weeks)
  * 5-FU bolus + infusions (400 mg/m^2) on days 1, 2, 15 and 16
  * Folinic Acid infusions (200 mg/m^2) on days 1, 2, 15 and 16
  Arms: 2

SUMMARY:
This is an exploratory study to compare activity and safety in 400 patients with previously untreated metastatic carcinoma of the colon treated with UFOX (a combination regimen of UFT® (Tegafur plus Uracil), Oxaliplatin, Folinic Acid) plus Cetuximab or FOLFOX-4 (a combination regimen of 5 Fluorouracil (5-FU), Oxaliplatin and Folinic Acid) plus Cetuximab)

ELIGIBILITY:
Inclusion Criteria

* Signed written informed consent
* Inpatient or outpatient ≥ 18 years of age
* Diagnosis of histologically confirmed adenocarcinoma of the colon or rectum
* First occurrence of metastatic disease (not curatively resectable)
* Presence of at least one lesion measurable uni dimensionally by computerised tomography (CT) scan or magnetic resonance imaging (MRI). (Target lesion(s) must not lie within an irradiated area)
* Life expectancy of ≥ 3 months
* Karnofsky performance status of ≥ 60, at study entry
* White blood cell count (WBC) ≥ 3 x 10^9/L, with neutrophils ≥ 1.5 x 10^9/L, platelets ≥ 100 x 10^9/L, and hemoglobin ≥ 9 g/dL
* Aspartate transaminase and alanine transaminase ≤ 2.5 x Upper Limit of Normal (ULN) (≤ 5 x ULN if liver metastasis are present)
* Normal serum creatinine (in case of elevated creatinine, labelled ethylenediaminetetraacetic acid clearance ≥ 65 mL/min is acceptable)
* Effective contraception for both male and female subjects if the risk of conception exists
* Tumor biopsy or archived sample available

Exclusion criteria:

* Brain metastasis and/or leptomeningeal disease (known or suspected)
* Previous chemotherapy for colorectal cancer except adjuvant treatment with progression of disease documented > 6 months after end of adjuvant treatment.
* Previous oxaliplatin-based chemotherapy
* Surgery (excluding diagnostic biopsy) or irradiation within 4 weeks prior to randomization
* Concurrent or previous chronic systemic immune therapy, targeted therapy, anti-vascular epithelial growth factor (VEGF) therapy, epidermal growth factor receptor (EGFR) pathway targeting therapy not indicated in the study protocol
* Concurrent hormonal therapy not indicated in the study protocol except for physiologic replacement or contraception
* Clinically relevant coronary artery disease, history of myocardial infarction in the last 12 months, or high risk of uncontrolled arrhythmia
* Peripheral neuropathy >grade 1
* Known hypersensitivity reaction to any of the components of the treatment.
* Any concurrent malignancy other than basal cell cancer of the skin, or pre-invasive cancer of the cervix. (Subjects with a previous malignancy but without evidence of disease for ≥ 5 years will be allowed to enter the study)
* Pregnancy (absence to be confirmed by ß-human chorionic gonadotrophin test) or lactation period
* Known drug abuse/alcohol abuse
* Legal incapacity or limited legal capacity
* Medical or psychological condition which in the opinion of the investigator would not permit the subject to complete the study or sign meaningful informed consent
* Participation in another clinical study within the 30 days before randomization
* Significant disease which, in the investigator's opinion, would exclude the subject from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2007-02; Primary Completion 2009-06 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Yves Douillard, MD PhD, Principal Investigator — Centre R Gauducheau
Locations (57):
- Argentina (2):
  - Research Site, Buenos Aires
  - Research Site, Ciudad Autónoma Buenos Aires
- Australia (2):
  - Research Site, Perth
  - Research Site, Wollongong
- Austria (2):
  - Research Site, Graz
  - Research Site, Vienna
- Belgium (2):
  - Research Site, Leuven
  - Research Site, Liège
- Brazil (3):
  - Research Site, Belo Horizonte
  - Research site, Cep Sao Paulo-SP
  - Research Site, Fortaleza
- France (8):
  - Research Site, Besançon
  - Research Site, Caen
  - Research Site, La Roche-sur-Yon
  - Research Site, Lille
  - Research Site, Marseille
  - Research Site, Nice
  - Research Site, Saint-Herblain
  - Research Site, Strasbourg
- Germany (13):
  - Research Site, Berlin
  - Research Site, Dortmund
  - Research Site, Dresden
  - Research Site, Frankfurt am Main
  - Research Site, Hamburg
  - Research Site, Hanover
  - Research Site, Heidelberg
  - Research Site, Kassel
  - Research Site, Krefeld
  - Research Site, Magdeburg
  - Research Site, München
  - Research Site, Oldenburg
  - Research Site, Wiesbaden
- Greece (3):
  - Research Site, Dragana
  - Research Site, Thessaloniki
  - Research Site, Voútai
- Hong Kong (2):
  - Research Site, Hong Kong
  - Research Site, Shatin
- Israel (2):
  - Research Site, Haifa
  - Research Site, Jerusalem
- Italy (11):
  - Research Site, Benevento
  - Research Site, Brescia
  - Research Site, Cremona
  - Research Site, Forlì
  - Research Site, Padua
  - Research Site, Pavia
  - Research Site, Potenza
  - Research Site, Reggio Emilia
  - Research Site, Rimini
  - Research Site, Roma
  - Research Site, Sassari
- Research Site, Mexico City, Mexico
- Poland (4):
  - Research Site, Krakow
  - Research Site, Lublin
  - Research Site, Opole
  - Research Site, Warsaw
- Thailand (2):
  - Research Site, Bangkok
  - Research Site, Pathumwan

REFERENCES:
- [Result] Douillard JY, Zemelka T, Fountzilas G, Barone C, Schlichting M, Heighway J, Eggleton SP, Srimuninnimit V. FOLFOX4 with cetuximab vs. UFOX with cetuximab as first-line therapy in metastatic colorectal cancer: The randomized phase II FUTURE study. Clin Colorectal Cancer. 2014 Mar;13(1):14-26.e1. doi: 10.1016/j.clcc.2013.11.009. Epub 2013 Nov 16. PMID 24370353

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject randomised 12 February 2007, last subject randomised 30 June 2008. Cut off date was 30th June 2009
Pre-assignment Details: A total of 329 participants were screened and 302 participants were included in the Intent to Treat (ITT) Population. One patient included in the ITT population received no study medication and was not included in the Safety Population which comprised 301 participants (151 received UFOX plus cetuximab and 150 FOLFOX4 plus cetuximab).
Groups:
- UFOX + Cetuximab: UFOX is a combination regimen of UFT® (Tegafur plus Uracil), Oxaliplatin and Folinic Acid.
  * Cetuximab infusion (400 mg/m^2 on day 1 of cycle 1 and 250 mg/m^2 at each subsequent day 1, as well as on days 8, 15 and 22)
  * Oxaliplatin infusion (85mg/m^2) on days 1 and 15 (every 2 weeks)
  * Oral UFT® (250mg/m^2 tegafur + 560 mg/m^2 uracil in 3 daily doses rounded to the nearest number of whole capsules) on days 1-21
  * Oral Folinic Acid (90 mg in 3 daily divided doses) on days 1-21
- FOLFOX4 + Cetuximab: FOLFOX4 is a combination regimen of 5 Fluorouracil (5-FU), Oxaliplatin and Folinic Acid.
  * Cetuximab infusion (400 mg/m^2 on day 1 of cycle 1 and 250 mg/m^2 at each subsequent day 1, as well as on days 8, 15 and 22)
  * Oxaliplatin infusion (85 mg/m^2) on days 1 and 15 (every 2 weeks)
  * 5-FU bolus + infusions (400 mg/m^2) on days 1, 2, 15 and 16
  * Folinic Acid infusions (200 mg/m^2) on days 1, 2, 15 and 16
Period: Overall Study
Arm/Group | UFOX + Cetuximab | FOLFOX4 + Cetuximab
Started | 152 | 150
Completed | 150 | 150
Not Completed | 2 | 0
Not completed — Subject on treatment | 1 | 0
Not completed — Subject in survival follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | UFOX + Cetuximab | FOLFOX4 + Cetuximab | Total
Number analyzed (Participants) | 152 | 150 | 302
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.1 (10.01) | 61 (11.04) | 60.5 (10.53)
Age, Customized [Number; unit: participants]
  <65 years | 93 | 84 | 177
  >=65 years | 57 | 66 | 123
  Missing | 2 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 55 | 112
  Male | 95 | 95 | 190
Region of Enrollment [Number; unit: participants]
  Hong Kong | 7 | 4 | 11
  Greece | 9 | 5 | 14
  Thailand | 7 | 9 | 16
  Austria | 13 | 9 | 22
  Italy | 28 | 33 | 61
  France | 6 | 8 | 14
  Mexico | 4 | 0 | 4
  Argentina | 5 | 6 | 11
  Brazil | 5 | 9 | 14
  Poland | 30 | 27 | 57
  Belgium | 5 | 7 | 12
  Australia | 6 | 5 | 11
  Germany | 27 | 28 | 55

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: Duration from randomization until progression or death due to any cause. Only deaths within 12 weeks of last tumor assessment are considered. Patients without event are censored on the date of last tumor assessment. Response and progression were assessed by the Investigators using response evaluation criteria in solid tumors (RECIST) 1.0 criteria
Time Frame: Time from randomization to disease progression, death, or last tumor assessment reported between day of first patient randomised, Feb 2007, until cut off date, 30 Jun 2009
Population: Intention-to-treat (ITT) population i.e. all randomized subjects .
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | UFOX + Cetuximab | FOLFOX4 + Cetuximab
Number analyzed (Participants) | 152 | 150
months | 6.6 [5.6 to 7.2] | 8.2 [7.5 to 9.2]
Statistical Analysis 1: Comparison: UFOX + Cetuximab vs FOLFOX4 + Cetuximab; Test type: Superiority or Other; p = 0.0048, Stratified log rank; Kaplan-Meier method was used to estimate median PFS time. HR was calculated using Cox proportional hazards model stratified by randomization strata; Hazard Ratio (HR) = 0.677, 95% CI 2-sided [0.515 to 0.889]

2. Secondary Outcome: Best Overall Response (BOR)
Description: BOR defined as percentage of subjects, whose BOR was either (confirmed) complete response (CR) or partial response (PR), relative to the number of subjects belonging to the study population of interest. CR defined as "Disappearance of all target lesions plus disappearance of all non-target lesions & without appearance of any new lesions; confirmed minimum 4 weeks later. PR defined as "At least 30% reduction in the SOLD of target lesions plus no significant change in non-target lesions to qualify for either CR or PD without appearance of new lesions; confirmed minimum 4 weeks later
Time Frame: Evaluations were performed every 8 weeks until disease progression, reported between day of first patient randomised, Feb 2007, until cut off date, 30 Jun 2009
Population: ITT population i.e. all randomized subjects.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | UFOX + Cetuximab | FOLFOX4 + Cetuximab
Number analyzed (Participants) | 152 | 150
percentage of participants | 37.5 [29.8 to 45.7] | 51.3 [43.0 to 59.6]
Statistical Analysis 1: Comparison: UFOX + Cetuximab vs FOLFOX4 + Cetuximab; Test type: Superiority or Other; p = 0.016, Cochran-Mantel-Haenszel; Stratified odds ratio and Cochran-Mantel- Haenszel (CMH) statistics were calculated considering the randomization strata; Odds Ratio (OR) = 1.756, 95% CI 2-sided [1.110 to 2.777]

3. Secondary Outcome: Overall Survival (OS)
Description: Time from randomization to death. Patients without event are censored at the last date known to be alive or at the clinical cut-off date, whatever is earlier.
Time Frame: Time from randomization to death or last known to be alive, reported between day of first patient randomised, Feb 2007, until cut off date, 30 Jun 2009
Population: ITT population i.e. all randomized subjects.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | UFOX + Cetuximab | FOLFOX4 + Cetuximab
Number analyzed (Participants) | 152 | 150
months | 12.9 [11.5 to 15.8] | 15.5 [12.6 to 18.1]
Statistical Analysis 1: Comparison: UFOX + Cetuximab vs FOLFOX4 + Cetuximab; Test type: Superiority or Other; p = 0.3797, Stratified log rank; Kaplan-Meier method was used to estimate median OS time. HR was calculated using Cox proportional hazards model stratified by randomization strata; Hazard Ratio (HR) = 0.855, 95% CI 2-sided [0.603 to 1.213]

4. Secondary Outcome: Overall Survival (OS)
Description: as for outcome 3
Time Frame: Time from randomization to death or last known to be alive, reported between day of first patient randomised, Feb 2007, until cut off date, 31 Aug 2011
Population: ITT population i.e. all randomized subjects.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | UFOX + Cetuximab | FOLFOX4 + Cetuximab
Number analyzed (Participants) | 152 | 150
months | 16.8 [13.9 to 18.5] | 18.4 [15.3 to 20.9]
Statistical Analysis 1: Comparison: UFOX + Cetuximab vs FOLFOX4 + Cetuximab; Test type: Superiority or Other; p = 0.8575, Stratified log rank; Hazard Ratio (HR) = 0.977, 95% CI 2-sided [0.755 to 1.263] — Kaplan-Meier method was used to estimate median OS time. HR was calculated using Cox proportional hazards model stratified by randomization strata

5. Secondary Outcome: Quality of Life (QOL) Functional Assessment of Cancer Therapy-Colorectal (FACT-C)
Description: All of the single-item measures of the FACT-C are assessed on ordinal response categories ranging from 0="Not at all" to 4="Very much". For scoring purposes the response scores are reversed on negatively phrased questions. The principle for scoring the sub-scales is the same in all cases: subscale score = (Sum of items × Number of items in the subscale) / numbers of items answered. The lowest possible total score is 0 and the highest is 136. A high scale score represents a high QOL.
Time Frame: At baseline, at every first day of every third cycle during active - treatment, and at final tumor assessment , reported between day of first patient randomised, Feb 2007, until cut-off date, 30 Jun 2009. Cycles were 4 weeks long unless dosing delays
Population: Patients were considered evaluable for FACT-C provided they had at least one evaluable FACT-C questionnaire and provided that they were also included in the ITT Population
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | UFOX + Cetuximab | FOLFOX4 + Cetuximab
Number analyzed (Participants) | 137 | 132
scores on a scale
  Baseline | 98.22 (1.725) | 96.45 (1.749)
  Cycle 3 | 95.41 (1.735) | 95.89 (1.806)
  Cycle 6 | 94.75 (2.090) | 94.70 (2.126)

6. Secondary Outcome: QOL EuroQuol-5D (EQ-5D) Health Outcome Questionnaire
Description: The EQ-5D questionnaire is a measure of health status that provides a simple descriptive profile and a single index value. The optional part of the questionnaire was not applied. The EQ-5D defines health in terms of mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The 5 items are combined to generate health profiles. These profiles were converted to a continuous single index score using a one to one matching. The lowest possible score is -0.59 and the highest is 1.00, higher scores on the EQ-5D represent a better QOL.
Time Frame: at baseline, at every first day of every third cycle during active - treatment, and at final tumor assessment , reported between day of first patient randomised, Feb 2007, until cut-off date, 30 Jun 2009. All cycles were 4 weeks long unless dosing delays
Population: Patients were considered evaluable for EQ-5D provided they had at least one evaluable EQ-5D questionnaire and provided that they were also included in the ITT Population.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | UFOX + Cetuximab | FOLFOX4 + Cetuximab
Number analyzed (Participants) | 136 | 130
scores on a scale
  Baseline | 0.747 (0.021) | 0.734 (0.021)
  Cycle 3 | 0.782 (0.021) | 0.758 (0.022)
  Cycle 6 | 0.758 (0.026) | 0.771 (0.026)

7. Secondary Outcome: QOL Therapy Preference Questionnaire (TPQ)
Description: TPQ was used to investigate which features of chemotherapy treatment are the most relevant in ensuring patient satisfaction. The most essential characteristics of a cancer medication are shown at baseline and at cycle 3, along with percentage of subjects selecting that characteristic.
Time Frame: as for outcome 6
Population: Patients were considered evaluable for TPQ provided they had at least one evaluable TPQ questionnaire and they were also included in the ITT TPQ subset population.
  The most essential characteristics of a cancer medication score are shown at baseline and cycle 3, no further cycles are available due to the low number of patients in later cycles
Measure: Number; unit: percentage of participants
Arm/Group | UFOX + Cetuximab | FOLFOX4 + Cetuximab
Number analyzed (Participants) | 99 | 99
percentage of participants
  Baseline: Does not increase your risk of infection | 18 | 16
  Baseline: Does not interfere with daily activities | 17 | 15
  Baseline: Does not make you vomit | 4 | 14
  Baseline: Does not give you diarrhea | 9 | 5
  Cycle 3: Does not increase your risk of infection | 15 | 15
  Cycle 3: Does not interfere with daily activities | 10 | 11
  Cycle 3: Does not make you vomit | 4 | 10
  Cycle 3: Does not give you diarrhea | 15 | 4

8. Secondary Outcome: Treatment Impact on Social Daily Living and Health Care Resource Utilization
Description: Non-protocol medical care visits and consultations
Time Frame: From randomisation until final visit, reported between day of first patient randomised, Feb 2007, until cut-off date, 30 Jun 2009
Population: ITT population
Measure: Number; unit: visits or consultations
Arm/Group | UFOX + Cetuximab | FOLFOX4 + Cetuximab
Number analyzed (Participants) | 152 | 150
visits or consultations
  Emergency room visit | 34 | 26
  Hospital oupatient clinic visit | 40 | 35
  Practice visit | 71 | 159
  Home visit | 15 | 130
  General Practitioner consultation | 65 | 124
  Specialist consultation | 62 | 84
  Nurse consultation | 15 | 123
  Other consultation | 19 | 18

9. Secondary Outcome: Safety - Number of Patients Experiencing Any Adverse Event
Description: Please refer to Adverse Events section for details of individual serious adverse events and other adverse events
Time Frame: Time from first dose up to 30 days after last dose of study treatment, reported between day of first patient randomised, Feb 2007, until cut off date, 30 Jun 2009
Population: Safety population
Measure: Number; unit: participants
Arm/Group | UFOX + Cetuximab | FOLFOX4 + Cetuximab
Number analyzed (Participants) | 151 | 150
participants | 151 | 149

ADVERSE EVENTS:
Time Frame: Time from first dose up to 30 days after last dose of study treatment, reported between day of first patient randomised, Dec 2006, until cut off date, 30 Jun 2009
Arm/Group | UFOX + Cetuximab | FOLFOX4 + Cetuximab
Serious Adverse Events (participants affected / at risk) | 52/151 | 48/150
Other Adverse Events (participants affected / at risk) | 151/151 | 146/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | UFOX + Cetuximab (N=151) | FOLFOX4 + Cetuximab (N=150)
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 2
Splenic vein thrombosis (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Ulcerative keratitis (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 5 | 4
Anal fistula (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 13 | 4
Faecaloma (Gastrointestinal disorders) | 0 | 1
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 5 | 2
Intestinal obstruction (Gastrointestinal disorders) | 5 | 2
Nausea (Gastrointestinal disorders) | 4 | 0
Proctalgia (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1
Subileus (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 9 | 3
Asthenia (General disorders) | 0 | 1
Chills (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 2
General physical health deterioration (General disorders) | 0 | 4
Inflammation (General disorders) | 1 | 0
Pyrexia (General disorders) | 3 | 8
Biliary colic (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Hepatorenal syndrome (Hepatobiliary disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 2
Anal abscess (Infections and infestations) | 1 | 0
Catheter related infection (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Central line infection (Infections and infestations) | 1 | 5
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Hepatitis C (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1
Pyelonephritis (Infections and infestations) | 0 | 1
Pyelonephritis acute (Infections and infestations) | 1 | 0
Rectal abscess (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 1 | 2
Urinary tract infection (Infections and infestations) | 0 | 2
Urosepsis (Infections and infestations) | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 2
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Blood glucose abnormal (Investigations) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 1
Coma hepatic (Nervous system disorders) | 1 | 0
Grand mal convulsion (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 2
Anxiety (Psychiatric disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0
Ureteric perforation (Renal and urinary disorders) | 0 | 1
Urethral disorder (Renal and urinary disorders) | 1 | 0
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Vaginal fistula (Reproductive system and breast disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 0
Arterial thrombosis (Vascular disorders) | 0 | 1
Circulatory collapse (Vascular disorders) | 0 | 1
Femoral artery embolism (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | UFOX + Cetuximab (N=151) | FOLFOX4 + Cetuximab (N=150)
Neutropenia (Blood and lymphatic system disorders) | 10 | 65
Thrombocytopenia (Blood and lymphatic system disorders) | 33 | 37
Leukopenia (Blood and lymphatic system disorders) | 5 | 28
Anaemia (Blood and lymphatic system disorders) | 15 | 26
Conjunctivitis (Eye disorders) | 14 | 14
Diarrhoea (Gastrointestinal disorders) | 79 | 72
Nausea (Gastrointestinal disorders) | 67 | 55
Stomatitis (Gastrointestinal disorders) | 15 | 36
Vomiting (Gastrointestinal disorders) | 40 | 32
Constipation (Gastrointestinal disorders) | 29 | 30
Abdominal pain (Gastrointestinal disorders) | 34 | 25
Abdominal pain upper (Gastrointestinal disorders) | 10 | 8
Dyspepsia (Gastrointestinal disorders) | 10 | 8
Flatulence (Gastrointestinal disorders) | 9 | 1
Fatigue (General disorders) | 38 | 38
Pyrexia (General disorders) | 30 | 36
Mucosal inflammation (General disorders) | 15 | 34
Asthenia (General disorders) | 25 | 27
Oedema peripheral (General disorders) | 11 | 11
Chills (General disorders) | 5 | 9
Hyperbilirubinaemia (Hepatobiliary disorders) | 12 | 6
Drug hypersensitivity (Immune system disorders) | 12 | 10
Hypersensitivity (Immune system disorders) | 3 | 8
Paronychia (Infections and infestations) | 26 | 33
Folliculitis (Infections and infestations) | 8 | 14
Nasopharyngitis (Infections and infestations) | 6 | 11
Pharyngitis (Infections and infestations) | 8 | 7
Weight decreased (Investigations) | 12 | 16
Alanine aminotransferase increased (Investigations) | 9 | 8
Platelet count decreased (Investigations) | 9 | 6
Aspartate aminotransferase increased (Investigations) | 10 | 5
Anorexia (Metabolism and nutrition disorders) | 40 | 36
Hypokalaemia (Metabolism and nutrition disorders) | 17 | 15
Hypomagnesaemia (Metabolism and nutrition disorders) | 15 | 14
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 10
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 8
Paraesthesia (Nervous system disorders) | 38 | 43
Peripheral sensory neuropathy (Nervous system disorders) | 29 | 27
Neuropathy peripheral (Nervous system disorders) | 17 | 22
Dysgeusia (Nervous system disorders) | 13 | 20
Polyneuropathy (Nervous system disorders) | 6 | 17
Headache (Nervous system disorders) | 6 | 10
Dysaesthesia (Nervous system disorders) | 11 | 5
Insomnia (Psychiatric disorders) | 9 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9 | 13
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 7
Rash (Skin and subcutaneous tissue disorders) | 63 | 47
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 40 | 45
Dry skin (Skin and subcutaneous tissue disorders) | 27 | 29
Skin fissures (Skin and subcutaneous tissue disorders) | 13 | 22
Pruritus (Skin and subcutaneous tissue disorders) | 8 | 15
Acne (Skin and subcutaneous tissue disorders) | 20 | 14
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 10 | 13
Alopecia (Skin and subcutaneous tissue disorders) | 6 | 13
Erythema (Skin and subcutaneous tissue disorders) | 10 | 12
Nail disorder (Skin and subcutaneous tissue disorders) | 7 | 11
Dermatitis (Skin and subcutaneous tissue disorders) | 5 | 9
Hypertension (Vascular disorders) | 8 | 11

LIMITATIONS AND CAVEATS:
Dosing of UFT/ folinic acid in the experimental arm were not directly recorded, so dosing data is not fully available in the UFOX plus cetuximab arm (36/151). Comparative conclusions on drug exposure might be impacted by a bias due to missing data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other